CLINICAL TRIAL: NCT05524883
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study Assessing Safety, Tolerability, Pharmacodynamics, Efficacy, and Pharmacokinetics of DYNE-251 Administered to Participants With Duchenne Muscular Dystrophy Amenable to Exon 51 Skipping
Brief Title: Safety, Tolerability, Pharmacodynamic, Efficacy, and Pharmacokinetic Study of DYNE-251 in Participants With Duchenne Muscular Dystrophy Amenable to Exon 51 Skipping
Acronym: DELIVER
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dyne Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DYNE251-DMD-201; 2023-510351-31-00 (EU CTIS Number); ITA 362546 (model PA-000798) (Other: Health Canada Investigational Testing Authorization (ITA))
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo-Controlled MAD Period - DYNE-251 (Experimental): DYNE-251 will be administered once every 4 weeks (Q4W) or once every 8 weeks (Q8W) over 24 weeks.
  Interventions: Drug: DYNE-251
- Placebo-Controlled MAD Period - Placebo (Experimental): Placebo will be administered Q4W or Q8W over 24 weeks.
  Interventions: Drug: Placebo
- Open-Label and Long-Term Extension Period - DYNE-251 (Experimental): DYNE-251 will be administered Q4W or Q8W for up to 192 weeks after participants complete the Placebo-Controlled MAD Period of the study.
  Interventions: Drug: DYNE-251

INTERVENTIONS:
Drug: DYNE-251 — Administered by IV infusion
  Arms: Open-Label and Long-Term Extension Period - DYNE-251; Placebo-Controlled MAD Period - DYNE-251
Drug: Placebo — Administered by IV infusion
  Arms: Placebo-Controlled MAD Period - Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, and dystrophin protein levels in muscle tissue following multiple intravenous (IV) doses of DYNE-251 in participants with Duchenne muscular dystrophy (DMD) amenable to exon 51 skipping.

The study consists of 3 periods: a multiple-ascending dose (MAD) / placebo-controlled period (24 weeks), an open-label period (24 weeks) and a long-term extension (LTE) period (192 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 16 years inclusive, at the time of informed consent/assent.
* Male with a confirmed diagnosis of DMD and with a mutation in the dystrophin gene characterized by exon deletion amenable to exon 51 skipping.
* Upper extremity muscle group that is amenable to muscle biopsy.
* Brooke Upper Extremity Scale score of 1 or 2.
* Ambulatory or non-ambulatory. A non-ambulatory participant must have been non-ambulatory for <2 years before enrollment.
* Receiving a stable dosage of glucocorticoids for at least 12 weeks prior to the start of study drug administration, with the expectation of maintaining a stable dose during the Placebo-Controlled and Open-Label Periods of the study (unless dose adjustment is required by weight change).
* Left ventricular ejection fraction of ≥50% by echocardiogram or ≥55% by cardiac magnetic resonance imaging (MRI).

Exclusion Criteria:

* Uncontrolled clinical symptoms and signs of congestive heart failure (CHF).
* Any change in prophylaxis/treatment for CHF within 3 months prior to the start of study treatment.
* History of major surgical procedure within 12 weeks prior to the start of study drug administration or an expectation of a major surgical procedure during the study.
* Requirement of daytime ventilator assistance.
* Percent predicted FVC <40 % (applies only for participants who are age ≥7 years).
* Receipt of eteplirsen, or alternative exon-skipping/dystrophin-modifying therapy, within 12 weeks of randomization.
* Receipt of non-exon skipping investigational drug within 4 months before the start of study drug administration.
* Receipt of gene therapy at any time.

Other inclusion and exclusion criteria may apply.

Ages: 4 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 86 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Through study completion, up to Week 241
Change From Baseline in Dystrophin Protein Levels in Muscle Tissue at Week 25 | Baseline, Week 25

SECONDARY OUTCOMES:
Change From Baseline in Muscle Tissue Exon 51 Skipping Levels at Week 25 For Participants Dosed at Q4W or Q8W Interval With a Second Biopsy Performed at Week 25 | Baseline, Week 25
Change From Baseline in Muscle Tissue Percent Dystrophin-Positive Fiber (PDPF) at Week 25 For Participants Dosed at Q4W or Q8W Interval With a Second Biopsy Performed at Week 25 | Baseline, Week 25
Change From Baseline in Blood Creatine Kinase (CK) Levels up to Week 241 For Participants Dosed at Q4W or Q8W Interval With a Second Biopsy Performed at Week 25 | Baseline, up to Week 241
Change From Baseline in Dystrophin Protein Level in Muscle Tissue as Determined by Western Blot at Week 49 For Participants Dosed at Q8W Interval With a Second Biopsy Performed at Week 49 | Baseline, Week 49
Change From Baseline in Muscle Tissue Exon 51 Skipping Levels at Week 49 For Participants Dosed at Q8W Interval With a Second Biopsy Performed at Week 49 | Baseline, Week 49
Change From Baseline in Muscle Tissue PDPF at Week 49 For Participants Dosed at Q8W Interval With a Second Biopsy Performed at Week 49 | Baseline, Week 49
Change From Baseline in Blood CK Levels up to Week 241 For Participants Dosed at Q8W Interval With a Second Biopsy Performed at Week 49 | Baseline, up to Week 241
Change From Baseline in North Star Ambulatory Assessment (NSAA) Total Score in Ambulatory Participants up to Week 241 | Baseline, up to Week 241
  The NSAA is a 17-item functional scale used to measure functional motor abilities in ambulant participants with DMD and monitor progression of the disease and treatment effects in each of the items. The items are graded on a 3-point scale: 0=unable to achieve independently, 1=modified method but achieves goal with no physical assistance, and 2=normal, no obvious modification of activity. Total score range is 0 to 34.
Change From Baseline in Time to Rise From Floor in Ambulatory Participants up to Week 241 | Baseline, up to Week 241
Change From Baseline in 10-Meter Run/Walk (10MRW) Time in Ambulatory Participants up to Week 241 | Baseline, up to Week 241
Change From Baseline in Performance Upper Limb (PUL) Scale Version 2.0 Score up to Week 241 | Baseline, up to Week 241
  The PUL scale is a validated tool specifically designed for assessing upper limb function in ambulant and non-ambulant individuals with DMD. It includes an entry item to define the broad starting functional level and 22 items subdivided into 3 areas indicative of upper limb strength as, shoulder level, midlevel, and distal level. The global score is a combination of the 3 areas and ranges from 0 to 42. Lower scores indicate higher disability.
Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) up to Week 241 | Baseline, up to Week 241
Change From Baseline in Stride Velocity 95th Centile (SV95C) in Ambulatory Participants up to Week 241 | Baseline, up to Week 241
Maximum Observed Plasma Drug Concentration of DYNE-251 (Cmax) | Through study completion, up to Week 241
Time to Maximum Observed Plasma Drug Concentration of DYNE-251 (tmax) | Through study completion, up to Week 241
Area Under the Plasma Drug Concentration-Time Curve From Time 0 to the Last Quantifiable Concentration of DYNE-251 in Plasma (AUC0-tlast) | Through study completion, up to Week 241
Area Under the Plasma Drug Concentration Versus Time Curve From Time 0 (Dosing) Extrapolated to Time Infinity of DYNE-251 (AUC∞) | Through study completion, up to Week 241
Apparent Terminal Phase Elimination Rate Constant of DYNE-251 in Plasma (λz) | Through study completion, up to Week 241
Apparent Terminal Elimination Half-Life of DYNE-251 in Plasma (t½) | Through study completion, up to Week 241
Total Body Clearance (CL) of DYNE-251 | Through study completion, up to Week 241
Volume of Distribution at the Terminal Phase of DYNE-251 in Plasma (Vz) | Through study completion, up to Week 241
Volume of Distribution at Steady State of DYNE-251 in Plasma (Vss) | Through study completion, up to Week 241
Tissue Phosphorodiamidate Morpholino Oligomer (PMO) Concentration of DYNE-251 in Muscle Tissue | Through study completion, up to Week 241
Percentage of Participants With Antidrug Antibodies (ADAs) | Through study completion, up to Week 241

CONTACTS AND LOCATIONS:
Locations (30):
- United States (11):
  - University of California San Diego, La Jolla, California
  - UCLA University California of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rare Disease Research, LLC, Atlanta, Georgia
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio
  - Shriners Hospitals for Children Portland, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah - PPDS, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Murdoch Children's Research Institute, Parkville, Victoria
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHR Citadelle, Liège
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
- CHI [Children's Health Ireland] at Temple Street Children's University Hospital, Dublin, Ireland
- Italy (3):
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Fondazione Serena Onlus - Centro Clinico NeMO, Milan, Lombardy
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
- Samsung Medical Center, Seoul, Teugbyeolsi, South Korea
- Spain (2):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Sant Joan de Déu Universidad de Barcelona, Barcelona
- United Kingdom (5):
  - Alder Hey Children's Hospital, Liverpool, Merseyside
  - Royal Victoria Infirmary, Newcastle upon Tyne, Northumberland
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - Bristol Childrens Hospital, Bristol
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: No